CLINICAL TRIAL: NCT02834130
Title: Input of a Multidisciplinary Device Including a Psychological Approach, to Accompany the Announce of Diagnosis for Young Children With Serious Constitutional Hemorrhagic Disease and Their Families
Brief Title: Input of a Multidisciplinary Device to Accompany the Announce of Diagnosis for Young Children With Serious Constitutional Hemorrhagic Disease and Their Families
Acronym: ACADHEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-05; 2014-A00367-40 (Registry Identifier: Ansm)
Record Dates: First submitted 2015-10-21; First posted 2016-07-15 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Severe Forms of Hemophilia; Other Constitutional Bleeding Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- children from 2 to 10 years with haemophilia or allied HBD, wh (Other)
  Interventions: Behavioral: Evaluation of psychological and psychopathological

INTERVENTIONS:
Behavioral: Evaluation of psychological and psychopathological
  Other Names: Evaluation of quality of life

SUMMARY:
Severe forms of hemophilia and other constitutional bleeding disorders represent a group of rare diseases. In last decades, news therapies have dramatically increased life expectancy and joint's protection.

The investigators propose to set up a single-centre, descriptive, transversal pilot study, designed for the inclusion of around thirty children from 2 to 10 years, with haemophilia or allied hereditary bleeding disorders (HBD), who were referred to the Hemophilia Treatment Center (HTC) of Marseille at diagnosis. For those children who were able to benefit from the totality or part of the device accompanying the diagnostic announcement in the past 10 years.

DETAILED DESCRIPTION:
Severe forms of hemophilia and other constitutional bleeding disorders represent a group of rare diseases. In last decades, news therapies have dramatically increased life expectancy and joint's protection. The recurrence of joint bleedings is responsive of multifocal arthropathy in the natural history, but nowadays, the orthopedic outcome is good thanks to prophylactic treatments.

However, the announcement of the diagnosis of such hereditary bleeding disorders at a very young age represents a real psychological trauma for parents. Such an announcement may induce some psycho-developmental impairment.

An innovative support has been implemented at the Hemophilia Treatment Center in Marseille, in conjunction with the French Hemophilia Society. This program is based on a multidisciplinary partnership that favors the psychological support and the reinsurance of the parents.

With Rare Diseases Foundation support, the investigators have initiated this pilot study that will include more than 20 patients with severe hemophilia or constitutional bleeding disorder, who benefit from the device. This descriptive, monocentric, interventional study will permit to describe the psychological status, the quality of life of patients and their parents, but also to evaluate the impact of the device on initiation and observance of treatments like Long Term Prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 3 and 12 years
* Patients diagnosed and treated at the Center until inclusion
* Patients with FVIII :C < 2% or with FIX :C <2% or with FVII:C <2% or with FXIII:C <2% or fibrinogen <0,2 g/l, or with type 3 von Willebrand diseases or Thrombasthenia of Glanzmann diseases.
* Patient who participate to multidisciplinary support and announcement of diagnosis device
* Voluntarily given fully informed written and signed consents obtained before any study-related procedures are conducted

Exclusion Criteria:

* Patient with other clotting disorder or disease.
* Patient diagnosed or treated in other centre
* Patient with psychiatric disorder or disease
* Patient with other severe chronic disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Exposure Days compared to the Number of Treatment Exposure days prescribed | 2 years
  Treatment Observance

SECONDARY OUTCOMES:
Assessment of patient's behavioral condition using the Child Behavior Check-list (CBCL) 1,5-5 | 2 Years
Assessment of the patient's body consciousness through the "CORP-R" test (french test of body mapping) | 2 years
Assessment of patient's quality of life using the "Kidscreen" questionnaire for children | 2 years
Assessment of the patient's parents' Qaulity of life through the Short Form Health Survey (SF-36) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hopital Enfants de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France